CLINICAL TRIAL: NCT06131047
Title: Effects of High Intensity Resistance Training With and Without Blood Flow Restriction on Quadriceps Strength, Power and Agility in ACL Reconstruction Among Volley Ball Players
Brief Title: High Intensity Resistance Training With and Without Blood Flow Restriction in ACL Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0442
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Resistance Training; Blood Flow Restriction Therapy; Anterior Cruciate Ligament Reconstruction; Volleyball
Keywords: High intensity resistance training; Blood Flow Restriction Traning; ACL reconstruction; Volley ball Players

STUDY DESIGN:
Intervention Model Description: Randomized Clinical trial
Who Masked: Outcomes Assessor
Masking Description: Asessor who will take readings is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Traditional Resistance Training Group (Experimental): Group A will undergo Traditional Resistance training without blood flow Restriction. A 30-minute progressive, weight training program will be initiated 8 weeks after the ACL-reconstruction and will be conducted subsequent to the individual based program. The resistance (training loads) will be increased when the individual could do more repetitions than the number specified in the weight training protocol. The exercises will be performed at a slow speed to ensure full control of the movement.
  Interventions: Other: High intensity Traditional Resistance Traning without Blood Flow Restriction
- High Intensity Traditional Resistance Training with Blood Flow Restriction Group (Experimental): Group B will perform low-load blood flow restriction (LL-BFR) training using external loads of 20-40% 1RM has been suggested as an alternative to traditional strength rehabilitation. Minimum of 2 -3 sets and maximum total 5 sets,20-30 repetitions of each exercise with 30 to 60 seconds rest period and 2-3 times per weekly for 4-6 weeks to During LL-BFR training, a pressurized cuff is applied to the proximal thigh that oc¬cludes venous outflow while maintaining arterial in¬flow. The combination of venous occlusion and resis¬tance training is believed to induce muscle hypertrophy secondary to elevated systematic hormone production, cell swelling, production of reactive oxygen species, intramus¬cular anabolic signaling and fast-twitch fiber recruit¬ment.(
  Interventions: Other: High intensity Traditional Resistance Traning with Blood Flow Restriction

INTERVENTIONS:
Other: High intensity Traditional Resistance Traning without Blood Flow Restriction — Group A will undergo Traditional Resistance training without blood flow Restriction. A 30-minute progressive, weight training program will be initiated 8 weeks after the ACL-reconstruction and will be conducted subsequent to the individual based program. The resistance (training loads) will be increased when the individual could do more repetitions than the number specified in the weight training protocol. The exercises will be performed at a slow speed to ensure full control of the movement
  Arms: High Intensity Traditional Resistance Training Group
Other: High intensity Traditional Resistance Traning with Blood Flow Restriction — Group B will recieve low-load blood flow restriction (LL-BFR) training using external loads of 20-40% 1RM has been suggested as an alternative to traditional strength rehabilitation. Minimum of 2 -3 sets and maximum total 5 sets,20-30 repetitions of each exercise with 30 to 60 seconds rest period and 2-3 times per weekly for 4-6 weeks to During LL-BFR training, a pressurized cuff is applied to the proximal thigh that oc¬cludes venous outflow while maintaining arterial in¬flow. The combination of venous occlusion and resis¬tance training is believed to induce muscle hypertrophy secondary to elevated systematic hormone production, cell swelling, production of reactive oxygen species, intramus¬cular anabolic signaling and fast-twitch fiber recruit¬ment
  Arms: High Intensity Traditional Resistance Training with Blood Flow Restriction Group

SUMMARY:
This study is randomized and single-blinded. Ethical approval is taken from the ethical committee of riphah international university, Lahore. Participants who meet the inclusion criteria will be enrolled in Groups A & B through the sealed envelop method by the Non-Probability Convenient random sampling technique. Group A will perform traditional High-intensity resistance training without Blood Flow Restriction training after ACL Reconstruction Surgery. Group B will perform traditional High-intensity Resistance training with Blood Flow Restriction training after ACL Reconstruction Surgery.

DETAILED DESCRIPTION:
The objective of the study is to determine the effects of high-intensity resistance training with and without blood flow restriction on quadriceps strength, power, and agility after ACL reconstruction among volleyball players. This study is randomized and single-blinded. Ethical approval is taken from the ethical committee of riphah international university, Lahore. Participants who meet the inclusion criteria will be enrolled in Groups A & B through the sealed envelop method by the Non-Probability Convenient random sampling technique. Group A will perform traditional High-intensity resistance training without Blood Flow Restriction training after ACL Reconstruction Surgery. Group B will perform traditional High-intensity Resistance training with Blood Flow Restriction training after ACL Reconstruction Surgery. The outcome measures will be assessed by hand held dynamometer.1-RM test, Illinois Agility Test, and Vertical jump test.

The data will be analyzed by SPSS,version 25.Statistical siginificance is P= 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Male players with age group 18 to 25 years,Return to function phase of rehabilitation,Players with Grade III ACL Tear ,Athletes who have been playing for at least 2 years

Exclusion Criteria:

* Players after ACL Reconstruction in acute or subacute phase,Players with other biomechanical issues of knee or feet,Players with any hematological disorders or hypertension

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Strength | Pre and 6 weeks post interventions
  strength will be measured with hand held dynamometer and 1-RM test
Agility | Pre and 6 weeks post interventions
  Illinois Agility Test Test will be used to measure agility
Power | Pre and 6 weeks post interventions
  Vertical Jump test will be used to measure power

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Nouman Tabassum, DPT, Principal Investigator — Ghurki Trust & Teaching Hospital,Lahore
Locations (1):
- Ghurki Trust & Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moses B, Orchard J, Orchard J. Systematic review: Annual incidence of ACL injury and surgery in various populations. Res Sports Med. 2012 Jul;20(3-4):157-79. doi: 10.1080/15438627.2012.680633. PMID 22742074
- [Background] Kruse LM, Gray B, Wright RW. Rehabilitation after anterior cruciate ligament reconstruction: a systematic review. J Bone Joint Surg Am. 2012 Oct 3;94(19):1737-48. doi: 10.2106/JBJS.K.01246. PMID 23032584
- [Background] Elabd OM, Elabd AM. Functional outcomes of a criterion-based rehabilitation protocol for anterior cruciate ligament reconstruction in amateur athletes: A randomised clinical trial. J Bodyw Mov Ther. 2023 Jul;35:7-13. doi: 10.1016/j.jbmt.2023.04.037. Epub 2023 Apr 17. PMID 37330806
- [Background] Kirby JC, Whitehead TS, Webster KE, Feller JA, McClelland JA, Klemm HJ, Devitt BM. Impact of Occupation on 12-Month Outcomes After Anterior Cruciate Ligament Reconstruction in Male Patients. Orthop J Sports Med. 2023 Feb 22;11(2):23259671221130377. doi: 10.1177/23259671221130377. eCollection 2023 Feb. PMID 36846817
- [Background] Lorenz DS, Bailey L, Wilk KE, Mangine RE, Head P, Grindstaff TL, Morrison S. Blood Flow Restriction Training. J Athl Train. 2021 Sep 1;56(9):937-944. doi: 10.4085/418-20. PMID 34530434
- [Background] Koc BB, Truyens A, Heymans MJLF, Jansen EJP, Schotanus MGM. Effect of Low-Load Blood Flow Restriction Training After Anterior Cruciate Ligament Reconstruction: A Systematic Review. Int J Sports Phys Ther. 2022 Apr 1;17(3):334-346. doi: 10.26603/001c.33151. eCollection 2022. PMID 35391871